CLINICAL TRIAL: NCT05113641
Title: Reducing Dietary Acid With Fruit and Vegetables Versus Oral Alkali in People With Chronic Kidney Disease (ReDACKD) Feasibility Trial
Brief Title: Reducing Dietary Acid With Food Versus Oral Alkali in People With Chronic Kidney Disease (ReDACKD)
Acronym: ReDACKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dylan MacKay (Other)
Collaborators: Dalhousie University (Other); Mount Saint Vincent University (Other)
Responsible Party: Sponsor-Investigator, Dylan MacKay, Assistant Professor, University of Manitoba
Organization: University of Manitoba (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS24768 (B2021:025)
Record Dates: First submitted 2021-10-15; First posted 2021-11-09 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Diseases; Metabolic Acidosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acidosis | interventions — Vegetables; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alkalizing Fruit and Vegetables (Experimental): Participants randomized to fruit and vegetables (F+V) will receive weekly supplementation of alkalizing fruits and vegetables via home delivery in a box format. Participants will receive a 1-hour dietary counseling session from a registered dietitian (RD), following randomization, either in person or via videoconference, depending on regional coronavirus disease (COVID) 19 restrictions and participant preference, which will outline the concepts of the dietary intervention. The RD will also recommend the best ways to prepare and include the F+V into the participant's current diet. Intervention will last 12 months.
  Interventions: Dietary Supplement: Alkalizing Fruit and Vegetables
- Sodium Bicarbonate (Active Comparator): Participants randomized to the alkali therapy will receive oral sodium bicarbonate 500mg tablets three times a day, reflecting a common starting dose at clinical practice. Thereafter, decisions around dose titration for the sodium bicarbonate will then be transferred to the participant's nephrologist who will be responsible for monitoring the participants serum bicarbonate concentration with a goal of maintaining a serum bicarbonate level >22 mEq/L. Participants will receive counselling from a registered dietician (RD) as part of the standard care. Intervention will last 12 months.
  Interventions: Drug: Sodium bicarbonate

INTERVENTIONS:
Dietary Supplement: Alkalizing Fruit and Vegetables — The weekly deliveries will contain combinations of fresh, frozen, and dried fruits and vegetables, as well as juices and soups which have been selected for their negative potential renal acid load (PRAL) values and shelf-life. All participants will be started at a F+V intake equal to -30 to -40 mEq per day reduction in dietary acid load estimated by the PRAL equation. Participants serum bicarbonate concentration will be measured at 1 month, and at 3 months, those with values < 22 mEq/L will have their recommended amount of F+V increased to -40 to -50 mEq per day. If a participant's 1- or 3-month serum bicarbonate value exceeds 29 mEq/L, their target dose of F+V in mEq/d will be reduced by 25%.
  Arms: Alkalizing Fruit and Vegetables
Drug: Sodium bicarbonate — Study nephrologist will prescribe the oral alkali therapy (sodium bicarbonate) and the medications will be dispensed by the dispensed by the clinic/hospital pharmacies.
  Arms: Sodium Bicarbonate

SUMMARY:
Metabolic acidosis is a common problem that occurs with worsening chronic kidney disease. Dietary acid can build up when the kidneys are not working well. This can be associated with a higher risk of worsening kidney function and death. The usual treatment is a medication called sodium bicarbonate which works to balance the acids in the body. The medication however often does not work and causes side effects. Consumption of alkalizing fruit and vegetables may work as a treatment for metabolic acidosis. This trial is being done to see if fruit and vegetables, provided via home delivery, can become a viable management for metabolic acidosis in patients with chronic kidney disease.

DETAILED DESCRIPTION:
Metabolic acidosis is a common complication of advanced chronic kidney disease (CKD). As kidney function declines, the ability to excrete excess dietary acid is reduced. This can lead to the development of metabolic acidosis, an imbalance in the body's acid-base balance. Metabolic acidosis is associated with a higher risk of CKD progression and mortality. Typical treatment includes an oral alkali, such as sodium citrate or sodium bicarbonate. Recent studies have shown that the treatment of metabolic acidosis can reduce the decline in kidney function and potentially prevent progression of CKD to dialysis. Treatment rates with an oral alkali are low because the treatments are ineffective, often poorly tolerated, and may be associated with net harm. Base producing fruit and vegetables are a potential treatment of metabolic acidosis by reducing the dietary contribution to overall acid load that must be managed by the kidneys. A recent systematic review and meta-analysis of clinical trials using oral alkali supplements or reduction in dietary acid intake using fruits and vegetables, when compared to no treatment, usual care or placebo found that these treatments increased serum bicarbonate and slowed the decline of kidney function. Fruit and vegetables are an effective and well-tolerated therapy for the treatment of metabolic acidosis in CKD. While oral alkali therapy has known adverse effects, important limitations also exist in the widespread applicability of fruit and vegetables as a treatment for metabolic acidosis. Only 2 single center randomized trials have examined the efficacy of fruit and vegetables for the management for acidosis. This dual-center trial will be the first randomized trial in Canada to evaluate the feasibility of providing fruit and vegetables via home delivery to patients for the management of metabolic acidosis in CKD. This study will be critical in designing a pan-Canadian phase 3 trial testing the efficacy of alkalizing fruit and vegetable provision on slowing the progression of CKD.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial
* Male or Female, aged 18 years or above
* Participants who have an eGFR between 15 and 40 ml/min/1.73m2
* Two consecutive measurements of serum bicarbonate of 14 to 22 mEq/L
* Systolic and diastolic blood pressure <160/100 mmHg
* Serum potassium <5.3 mmol/L
* Hemoglobin A1c below ≤ 11%
* Are registered in the nephrology clinic in Winnipeg or Halifax
* Participants are able to communicate in English and provide written informed consent

Exclusion Criteria:

* Anuria, dialysis or acute kidney injury/acute kidney failure in the 3 months prior to screening
* Chronic obstructive pulmonary disease that requires the participant to be on oxygen
* New York Heart Association Class 3-4 Heart failure symptoms or heart, liver or renal transplant
* A myocardial infarction or stroke within the last 6 months
* Unable to consume study treatments or control, such as swallowing or GI issues
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks
* Currently on potassium binding therapy
* Female participant who is pregnant or on lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Randomization to preliminary eligible ratio | 12 months
  Ratio of randomized to preliminary eligible greater, calculated among all patients approached to participate expressed as percentage will be collected at 12 months to investigate fruit and vegetable intervention feasibility.
  A red, yellow, green framework has been developed as a feasibility metric: green for ratios more than 50%, yellow for ratios 20%-49.9%, and red for ratios less than 20%
Weekly recruitment rate | 12 months
  Number of new participants per weeks of active recruitment. A green, yellow, red feasibility framework has been developed as a feasibility metric: green for ≥ 0.5 , yellow for 0.125-0.49 and red for < 0.125
Study outcome follow up | 12 months
  Study outcome follow up expressed as a percentage, will be calculated at 12 months to investigate the fruit and vegetable intervention feasibility. A red, yellow, green feasibility framework has been developed as a feasibility metric: green for ≥ 95% , yellow for 80%-94.9% and red for <80%.
Potential renal acid load (PRAL) in mEq/day | Baseline, 6, and 12 months
  Calculated from average dietary intake assessed by Automated Self-Administered 24-hour Canada (ASA24) dietary recall survey conducted over three days. a red, yellow, green feasibility framework has been developed as a feasibility metric: green for > 75% , yellow for 50%-75% and red for <50%.

SECONDARY OUTCOMES:
Five repetition chair stand time | Baseline, 3, 6, 9, and 12 months
  the amount of time it takes for a participant to get up out of a chair five times measured in seconds
Physical function related quality of life | Baseline, 3, 6, 9, and 12 months
  Participants will complete the SF-12 physical component score of the Kidney Disease Quality of Life Short Form (KDQOL-SF) questionnaire. The questionnaire is scored between 0-100 with higher values representing physical function related quality of life.
Serum bicarbonate (total CO2) | Baseline, 1, 3, 6, 9, and 12 month(s)
  Serum bicarbonate concentration in milliequivalents per liter (mEq/L)
Albumin | Baseline, 1, 3, 6, 9, and 12 month(s)
  blood albumin is measured in grams per deciliter (g/dL)
Calcium | Baseline, 1, 3, 6, 9, and 12 month(s)
  Total blood calcium concentration in mmol/L
Estimated Glomerular Filtration Rate (eGFR) | Baseline, 1, 3, 6, 9, and 12 month(s)
  calculated from serum creatinine, sex, and age, reported in mL/min/1.73 m2
Glucose | Baseline, 1, 3, 6, 9, and 12 month(s)
  Total blood glucose concentration in mmol/L
Potassium | Baseline, 1, 3, 6, 9, and 12 month(s)
  The total blood potassium concentration in mmol/L
Chloride | Baseline, 1, 3, 6, 9, and 12 month(s)
  Total blood chloride concentration in mmol/L
Sodium | Baseline, 1, 3, 6, 9, and 12 month(s)
  The total sodium concentration in mmol/L
Phosphorus | Baseline, 1, 3, 6, 9, and 12 month(s)
  The total blood phosphorus concentration in mmol/L
Hemoglobin A1c | Baseline, 1, 3, 6, 9, and 12 month(s)
  Hemoglobin A1c in percentage
Blood Urea Nitrogen (BUN) | Baseline, 1, 3, 6, 9, and 12 month(s)
  Blood Urea Nitrogen (BUN) is reported in millimole per litre (mmol/L)
Urine Albumin/Creatinine Ratio | Baseline, 1, 3, 6, 9, and 12 month(s)
  The ratio of albumin to creatinine concentrations in urine, reported in Milligrams albumin per millimole creatinine
Changes in medication | Baseline,1, 3, 6, 9, and 12 months
  Research coordinator will update information on concomitant medications or supplements information with the participant
Systolic blood pressure in mmHg | Baseline, 1, 3, 6, 9, and 12 months
  Blood pressure will be measured in triplicate using a validated blood pressure monitor following Kidney Disease: Improving Global Outcomes (KDIGO) 2021 measurement guidelines, the average of the 2nd and 3rd measurements will be recorded.
Diastolic blood pressure in mmHg | Baseline, 1, 3, 6, 9, and 12 months
  Blood pressure will be measured in triplicate using a validated blood pressure monitor following KDIGO 2021 measurement guidelines, the average of the 2nd and 3rd measurements will be recorded.
Edmonton Symptom Assessment System (ESAS) - Revised Renal | Baseline, 3, 6, 9, and 12 months
  A questionnaire used to rate the intensity of nine common symptoms experienced by renal patients, including pain, tiredness, drowsiness, nausea, appetite levels, shortness of breath, depression and anxiety levels, and well-being. Minimum value 0 and maximum value 100 with higher values being worse.
All cause hospitalization | 3, 6, 9, and 12 months
  Information on recent hospitalizations from participant's clinical records will be collected.
All cause mortality | 3, 6, 9, 12 months
  Information on mortality from participant's clinical records will be collected.
Height | Baseline, 3, 6, 9, and 12 months
  Height will be measured using a validated stadiometer in centimeters..
Weight | Baseline, 3, 6, 9, and 12 months
  Weight will be measured using a calibrated scale in kilograms.
Body Mass Index (BMI) | Baseline, 3, 6, 9, and 12 months
  MBI will be calculated through dividing weight in kilograms (kg) by the square of height in meters (m2).

OTHER OUTCOMES:
Exit Interviews | Final Visit (Month 12)-After the completion of the trial
  Upon the completion of the 12 months of study, the participants will be invited to participate in an exit interview. This interview will involve a few open ended question and its goal is to better understand participants' personal experiences and perspectives of the study and the intervention they received, as well as their overall viewpoints of trials such as ReDACKD, as a person living with CKD and metabolic acidosis. We will offer the interview to all of the participants at the final visit of the trial; however, taking part is this interview is voluntary.
  The "Exit Interview Consent Form" will be used to explain the aims and procedures of the interview

CONTACTS AND LOCATIONS:
Overall Officials: Navdeep Tangri, MD, PhD, Principal Investigator — Seven Oaks General Hospital Chronic Disease Innovation Centre; Dylan MacKay, PhD, Principal Investigator — George and Fay Yee Centre for Healthcare Innovation; Karthik Tennankore, MD, Principal Investigator — Nova Scotia Health Authority
Locations (3):
- Canada (3):
  - Seven Oaks General Hospital Chronic Disease Innovation Centre, Winnipeg, Manitoba
  - Health Sciences Center, Winnipeg, Manitoba
  - Chronic Kidney Disease (Renal) ClinicQEII - Dickson Building, Halifax, Nova Scotia

REFERENCES:
- [Derived] Mollard R, Cachero K, Luhovyy B, Martin H, Moisiuk S, Mahboobi S, Balshaw R, Collister D, Cahill L, Tennankore KK, Tangri N, MacKay D. Reducing Dietary Acid With Fruit and Vegetables Versus Oral Alkali in People With Chronic Kidney Disease (ReDACKD): A Clinical Research Protocol. Can J Kidney Health Dis. 2023 Aug 7;10:20543581231190180. doi: 10.1177/20543581231190180. eCollection 2023. PMID 37560749